CLINICAL TRIAL: NCT06583889
Title: Efficacy and Safety of endovasCular Treatment vs Standard Medical Care for Cerebral venOus Sinus thRombosis With mulTimodal Imaging Selection(ESCORT)
Brief Title: Endovascular Treatment or Standard Medical Care for Cerebral Venous Sinus Thrombosis(ESCORT)
Acronym: ESCORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dapeng Mo, Clinical Professor of Interventional Neuroradiology, Department of Neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YD2023001
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Venous Sinus Thrombosis
Keywords: Cerebral venous sinus thrombosis; Heparin; Randomized controlled trial; Endovascular treatment
MeSH Terms: interventions — Heparin; Tissue Plasminogen Activator; Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard medical care (Active Comparator)
  Interventions: Drug: Heparin
- Endovascular treatment with standard medical care (Experimental)
  Interventions: Procedure: Endovascular treatment

INTERVENTIONS:
Drug: Heparin — The patients randomized to standard medical care will receive (or continue) either any type of body-weight adjusted low molecular weight heparin in therapeutic dose, or intravenous adjusted dose unfractionated heparin (aPTT value kept within 1 time the normal value), according to the existing international guidelines.
  Arms: Standard medical care
Procedure: Endovascular treatment — Standard endovascular techniques to mechanically remove clot material, such as mechanical thrombectomy and/or balloon angioplasty and/or local application of alteplase or urokinase within the thrombosed sinuses.
  Other Names: Alteplase; Urokinase
  Arms: Endovascular treatment with standard medical care

SUMMARY:
Background: It has not been extensively studied in differing populations that endovascular treatment (EVT) for acute and subacute CVST with multimodal imaging selection improves the functional outcome better than standard medical care based on the guidelines. Published experience with endovascular treatment is promising. However, its efficacy has not been confirmed and early selection criteria for EVT are unknown.

Objective:The main objective of the Endovascular treatment or Standard medical Care for Cerebral Venous Sinus Thrombosis (ESCORT) trial is to determine if EVT improves the functional outcome of acute and subacute CVST patients with multimodal imaging selection.

Study Design:The ESCORT trial is a multicenter, prospective, randomized, open-label, blinded endpoint trial.

Study population: Patients are eligible if they have a radiologically criteria proven acute and subacute CVST, obvious symptoms of intracranial hypertension(lumbar puncture pressure≥250mmH2O).

Intervention: Patients will be randomized to receive either EVT or standard medical care (therapeutic doses of heparin). EVT consists of local application of alteplase or urokinase within the thrombosed sinuses, balloon angioplasty, and/or mechanical thrombectomy. Glasgow coma score, NIH stroke scale, ophthalmologic examination, Headache Impact Test-6(HIT-6), EuroQol-5 dimension-5 level(EQ-5D-5L) scale score, multimodal imaging and relevant laboratory parameters will be assessed at baseline.

Endpoints: The primary endpoint is the proportion with good prognosis at 3 months (definition: a. mRS≤1; b. headache score (<50, HIT-6); c. Frisén=0 grade for papilledema; d. defect of field vision PMD>-2dB). Secondary outcomes are three-months mRS, HIT-6,Frisén grade for papilledema, situation of EQ-5D-5L, mortality and recanalization rate. Major intracranial and extracranial hemorrhagic complications within one-week after the intervention are the principal safety outcomes. Results will be analyzed according to the'intention-to-treat' principle. Blinded assessors not involved in the treatment of the patient will assess endpoints with standardized questionnaires.

Study size: To detect a 20% relative increase of good prognosis (from 65 to 85%), 224 patients (112 in each treatment arm) have to be included (two-sided alpha, 80% power).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Included patients may benefit directly from EVT. Complications of EVT, most notably intracranial hemorrhages, constitute the most important risk of the study.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria

1. age between 18 years and 60 years
2. Cerebral venous sinus thrombosis (CVST), confirmed by computed tomographic and magnetic resonance imaging (T1, T2, SWI, DWI, FLAIR), magnetic resonance venography, computed tomographic venography or digital subtraction angiography.
3. Patients with CVST who meet the following conditions (1) Within 3 weeks of acute onset (2) There are one of the obvious clinical symptoms: A. symptoms of intracranial hypertension: headache, papilledema, visual acuity and visual field damage; B. Neurological impairment symptoms; C. Seizure; D. Disturbance of consciousness (GCS score≥9)
4. Lumbar puncture pressure≥250mmH2O
5. Patients or their relatives can sign written informed consent

Image inclusion criteria

1.CT and MRI (T1, T2, MRV, SWI, DWI) are used to screen CVST as acute phase (T1 low signal, T2 equal signal or slightly high signal; CT showed that the corresponding area is high signal) or subacute phase (T1 and T2 high signal) 2.3D-TOF or CE-MRA or CTV are used to screen the types of venous sinus thrombosis occlusion of main drainage which is prone to intracranial hypertension due to venous sinus thrombosis as follows: A.Superior sagittal sinus occlusion: thrombus obliterates the posterior 1/2 segment of superior sagittal sinus

B.Transverse sinus occlusive type:

1. complete thrombosis of the bilateral transverse sinus with or without the corresponding sigmoid sinus involvement
2. complete thrombosis of the superior transverse sinus with or without the corresponding sigmoid sinus involvement C.complete thrombosis of the superior sagittal sinus and unilateral transverse sinus with or without the corresponding sigmoid sinus involvement D.complete thrombosis of the superior sagittal sinus and bilateral transverse sinus with the corresponding sigmoid sinus is occluded

Exclusion Criteria:

1. Received any thrombolytic therapy within 7 days
2. Patients who cannot cooperate or accept MRI examination
3. Patients with dementia or mental illness are known to be unable to complete neurological function assessment and follow-up
4. Patients with high myopia and eye diseases affecting fundus examination and visual field examination
5. The patient has a clear history of primary headache such as migraine, tension headache and cluster headache, and a clear history of secondary headache
6. Patients who receive major surgery (excluding lumbar puncture) or a history of severe brain injury within 2 weeks
7. Known history of severe allergy to contrast media (excluding rash)
8. Gastrointestinal bleeding occurred within 3 months (excluding bleeding from recto anal hemorrhoids)
9. Serious liver function or renal dysfunction with written records and affecting normal coagulation function
10. Hemorrhagic disease (hemorrhagic disease history) with written records
11. Excepting for CVST, patients with any life expectancy less than 1 year (such as advanced cancer)
12. Pregnant women (puerperal women can be enrolled)
13. Patients with contraindications to anticoagulation or thrombolysis
14. Intracranial infectious or malignant tumor secondary to cerebrospinal fluid
15. CVST secondary to autoimmune diseases and hematological diseases (such as primary thrombocytosis, myelodysplastic syndrome, leukemia, etc.) and genetic factors
16. Concurrent thrombocytopenia (<100×109/L)
17. MRI features showed that the occluded vessels of venous sinus were in chronic phase (T1 and T2 images showed equal signal)
18. Severe brain tissue injury symptoms such as obvious space occupying effect due to massive cerebral edema, cerebral infarction or cerebral hemorrhage
19. Patients with CVST accompanied by ventricular compression and hydrocephalus requiring surgery
20. Participating in clinical trials of any other drugs or medical devices, or may participate in clinical trials of any other drugs or medical devices within 6 months after being enrolled in this clinical trial
21. The researchers judge that there are other situations that are not suitable for enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint | 90 days (±14 days) after randomization
  The proportion of good prognosis (definition: a. mRS≤1; b. headache score (<50, HIT-6); c. Frisén=0 grade for papilledema; d. defect of field vision PMD>-2dB)
Safety endpoint | Within 7 days after intervention treatment
  New intracranial hemorrhage or aggravation of intracranial hemorrhage after intervention treatment (including: symptomatic hemorrhage and all cerebral hemorrhage found by imaging. Symptomatic intracranial hemorrhage refers to any type of intracranial hemorrhage with NIHSS score increased by 4 points or more, even leading to death)
  Massive extracranial hemorrhage after intervention treatment (such as obvious clinical symptoms of extracranial organ system hemorrhage such as retroperitoneum, gastrointestinal tract, etc., accompanied by 2g/dl or more decrease in hemoglobin within 48 hours, or the need for infusion of 2 units or more of red blood cells, or the need for surgical intervention or even death)

SECONDARY OUTCOMES:
Favorable clinical outcome | 90 days (±14 days) after randomization
  mRS≤1
Headache Impact Test-6 (HIT-6) | 90 days (±14 days) after randomization
  HIT-6 score<50
Frisén grade for papilledema | 90 days (±14 days) after randomization
  The Frisén=0 grade
Perimetric Mean Deviation (PMD) | 90 days (±14 days) after randomization
  The perimetric mean deviation(PMD)>-2dB of visual field defect
Required surgical intervention in relation to CVST | within 90 days
  The proportion of surgical intervention within 90 days after randomization that are required in relation to cerebral venous thrombosis (e.g. ventricular shunting procedures or craniotomy)
Recanalization rate of cerebral venous sinus | 90 days (±14 days) after randomization
  The proportion of complete and partial recanalization of venous sinus (according to Qureshi classification criteria)
EuroQol-5 dimension-5 level(EQ-5D-5L) scale score | 90 days (±14 days) after randomization
All-cause mortality | 90 days after randomization
The incidence of cerebral hernia | 90 days after randomization
The proportion of decompressive craniectomy | 90 days after randomization
The incidence of other serious adverse events | 90 days after randomization

OTHER OUTCOMES:
The proportion of good prognosis | 12 months (±1 month) after randomization
  The proportion of good prognosis (defined as: a. mRS≤1, b. headache score (<50, HIT-6 score); c. Frisén grade=0 for papilledema; d. defect of field vision PMD>-2dB).
Favorable clinical outcome | 12 months (±1 month) after randomization
  mRS≤1
Headache Impact Test-6 (HIT-6) | 12 months (±1 month) after randomization
  HIT-6 score<50
Frisén grade for papilledema | 12 months (±1 month) after randomization
  The Frisén=0 grade
Perimetric Mean Deviation (PMD) | 12 months (±1 month) after randomization
  The perimetric mean deviation(PMD)>-2dB of visual field defect
Required surgical intervention in relation to CVST | 12 months (±1 month) after randomization
  The proportion of surgical intervention within 90 days after randomization that are required in relation to cerebral venous thrombosis (e.g. ventricular shunting procedures or craniotomy)
Recanalization rate of cerebral venous sinus | 12 months (±1 month) after randomization
  The proportion of complete and partial recanalization of venous sinus (according to Qureshi classification criteria)
Recurrence rate of venous sinus thrombosis | 12 months after randomization
EuroQol-5 dimension-5 level (EQ-5D-5L) scale score | 12 months (±1 month) after randomization
Interim analyses:good prognosis (definition: a. mRS≤1; b. headache score (<50, HIT-6); c. Frisén=0 grade for papilledema; d. defect of field vision PMD>-2dB) | After inclusion of 1/3rd and 2/3rd of patients
  The DSMB will perform two interim analyses after 75 and 150 patients (1/3rd and 2/3rd of all patients) have been randomized and completed the 12-month follow-up evaluation. As a stopping rule for efficacy, the Haybittle-Peto method will be used:1.Interim analysis 1: p=0,001;2.Interim analysis 2: p=0,001.In addition, the DSMB will assess futility during the interim analyses. The trial will be discontinued for futility if the conditional power is below 20%. This conditional power will be calculated under the assumption that in the remaining two-thirds/one-thirds of the study population the distributions of the primary endpoint will be the same as observed at the interim analysis.For theinterim analyses the DSMB will use the primary outcome measure (good prognosis: a. mRS≤1; b. headache score (<50, HIT-6); c. Frisén=0 grade for papilledema; d. defect of field vision PMD>-2dB at 12 months) for the determination of efficacy and futility.

CONTACTS AND LOCATIONS:
Overall Officials: Dapeng Mo, MD, Principal Investigator — Beijing Tiantan Hospital; Zhongrong Miao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No